CLINICAL TRIAL: NCT01383317
Title: Remote Ischemic Preconditioning (RIPC) and Its Effect on the Postoperative Pain Experience Following Intra-abdominal Surgery
Brief Title: Remote Ischemic PreConditioning Effect on Postsurgical Pain
Acronym: RIPCEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00016978
Record Dates: First submitted 2011-06-02; First posted 2011-06-28 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Remote Ischemic Preconditioning; Acute Pain
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RIPC (Active Comparator): A tourniquet on the thigh will be inflated to 300 mmHg for 5 minutes then deflated for 5 minutes. This will be repeated three times
  Interventions: Device: Thigh Tourniquet (VBM Single Use Tourniquet Cuff Items 20-34-722SLZ-1)
- Sham RIPC (Sham Comparator): A tourniquet on the thigh will be inflated to 15 mmHg for 5 minutes then deflated for 5 minutes. This will be repeated three times
  Interventions: Device: Sham RIPC

INTERVENTIONS:
Device: Thigh Tourniquet (VBM Single Use Tourniquet Cuff Items 20-34-722SLZ-1) — Disposable sterile thigh tourniquet
  Other Names: VBM Single Use Tourniquet Cuff Items 20-34-722SLZ-1
  Arms: RIPC
Device: Sham RIPC — Disposable sterile thigh tourniquet
  Other Names: VBM Single Use Tourniquet Cuff Items 20-34-722SLZ-1
  Arms: Sham RIPC

SUMMARY:
Remote Ischemic PreConditioning (RIPC) will improve the postoperative pain experience in patients undergoing abdominal surgery. Although abdominal surgery can be a lifesaving procedure many people have a significant amount of postsurgical pain. Severe postsurgical pain may lead to chronic pain in some people. "Remote Ischemic Preconditioning" may reduce the amount of postsurgical pain. Remote ischemic preconditioning is done by inflating a balloon (very similar to a blood pressure cuff) on the leg until it blocks blood flow for a few minutes. The cuff is then deflated and blood flow resumes. The process is repeated up to three times. This procedure causes the body to increase its natural pain relief system that may help to decrease the amount of postsurgical pain.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 30-80
2. Undergoing elective open intra-peritoneal surgery
3. Able to provide written informed consent to participate
4. Laparoscopic abdominal surgery

Exclusion Criteria:

1. Ongoing Workman's Compensation claim
2. >50mg/day of oral morphine or morphine equivalent
3. Currently being treated for lower extremity DVT
4. Known intracranial hypertension (not excluding patients with a functioning VP shunt)
5. Known Hypercoagulable state (e.g. factor V Leiden, protein s or c deficiency)
6. Ongoing localized thigh pain
7. Planned epidural analgesia
8. Pregnancy
9. Any DSM IV-R Axis I psychotic disorders
10. Unable to understand English
11. Unable to understand the consent form

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2016-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RIPC | Sham RIPC
Started | 29 | 35
Completed | 26 | 33
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIPC | Sham RIPC | Total
Number analyzed (Participants) | 29 | 35 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.03 (11.43) | 59.82 (10.62) | 55.52 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 10 | 12
  White | 23 | 18 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Pain Intensity and Unpleasantness Postoperatively
Description: Pain intensity and unpleasantness will be measured on postoperative day (POD) 1 and 2 by using a 0-10 verbal scale after asking the subject to cough. Higher scores denotes more intensity and unpleasantness of pain.
Time Frame: Postoperative day 1 and postoperative day 2
Population: Data was only collected for participants that were alert and conscious.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 19 | 23
units on a scale
  POD 1 | 4.82 (.71) | 4.83 (.62)
  POD 2 | 4.05 (3.08) | 4.81 (3.14)

2. Secondary Outcome: Number of Participants That Consumed Opioids
Description: All opioids administered during postoperative day (POD) 1 and 2 will be recorded and the number of participants that used opioids will be given.
Time Frame: Postoperative day 1 and postoperative day 2
Population: Data was not collected on some participants in both groups because they were unconscious, refused to answer or they were discharged.
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 25 | 25
Participants
  POD 1 | 20 | 24
  POD 2 | 19 | 22

3. Secondary Outcome: Consumption of Nonopioid Analgesics
Description: All non-opioids analgesics administered during postoperative day 1 and 2 will be recorded and the number of participants that used nonopiods will be given.
Time Frame: Postoperative day 1 and postoperative day 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 25 | 25
Participants
  POD 1 | 19 | 18
  POD 2 | 17 | 21

4. Secondary Outcome: Use of Antiemetics
Description: Number of participants that used an antiemetic postoperative day 1 and postoperative day 2 was recorded.
Time Frame: Postoperative day 1 and postoperative day 2
Population: Data was not collected on some participants in both groups because they were unconscious, refused to answer, or they were discharged.
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 25 | 23
Participants | 25 | 21

5. Secondary Outcome: Level of Sedation
Description: The Ramsey Sedation Scale (RSS) was used to determine the level of sedation. Th RSS defines the conscious state from a level 1: the patient is anxious, agitated or restless, through the continuum of sedation to a level 6: the patient is completely unresponsive. The score range is from 1-6, with higher scores denoting worse outcomes.
Time Frame: Postoperative day 1 and postoperative day 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 23 | 20
units on a scale
  POD 1 | 2.29 (.85) | 2.15 (.75)
  POD 2: number analyzed (Participants) | 20 | 20
  POD 2 | 2.11 (.65) | 1.95 (.39)

6. Secondary Outcome: McGill Pain Sensory
Description: The McGill Pain Questionnaire (MPQ) is a three-part pain assessment tool that measures several dimensions of the patient's pain experience. The scale range is 0-78, with higher scores denoting worse outcomes.
Time Frame: Postoperative day 1 and postoperative day 2
Population: Population differs from participant flow, because some participants in each group did not complete the assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 7 | 11
units on a scale
  POD 1 | 11.71 (9.36) | 12.73 (7.17)
  POD 2 | 7.14 (3.18) | 12.82 (12.21)

7. Secondary Outcome: Leg Pain at 48 Hours
Description: Number of participants that had leg pain at 48 hours.
Time Frame: postoperative day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 27 | 24
Participants | 4 | 1

8. Secondary Outcome: Patient Verbal Assessment as to Whether They Received Active Treatment or Placebo
Description: Participants were questioned to see if they knew what interventional group they belonged to.
Time Frame: Postoperative day 1 and postoperative day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 23 | 20
Participants
  Unsure/Unknown | 20 | 20
  RIPC | 1 | 0
  Sham | 2 | 0

9. Secondary Outcome: Pain Unpleasantness
Description: Pain unpleasantness will be measured on postoperative day (POD) 1 and 2 by using a 0-10 verbal scale after asking the subject to cough. Higher scores denotes more intensity and unpleasantness of pain.
Time Frame: Postoperative day 1 and postoperative day 2
Population: Data was not collected on some participants in both groups because they refused to answer or they were discharged.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RIPC | Sham RIPC
Number analyzed (Participants) | 19 | 25
units on a scale
  POD 1: number analyzed (Participants) | 19 | 24
  POD 1 | 4.43 (3.27) | 5.18 (3.7)
  POD 2: number analyzed (Participants) | 18 | 25
  POD 2 | 3.52 (3.46) | 4.54 (3.47)

ADVERSE EVENTS:
Arm/Group | RIPC | Sham RIPC
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes